CLINICAL TRIAL: NCT00333970
Title: Predictors of Response to Cognitive Remediation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F3460-V; JMF0001 (Other: VACHS)
Record Dates: First submitted 2006-06-02; First posted 2006-06-06 (Estimated); Results first posted 2014-10-09 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Schizophrenia
Keywords: cognition; neuropsychology; Rehabilitation; treatment efficacy; cognitive remediation
MeSH Terms: conditions — Schizophrenia | interventions — Cognitive Remediation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- cognitive remediation (Experimental): cognitive remediation
  Interventions: Behavioral: cognitive remediation
- treatment as usual (No Intervention): treatment as usual

INTERVENTIONS:
Behavioral: cognitive remediation — individual cognitive training
  Arms: cognitive remediation

SUMMARY:
The purpose of this study is to determine which variables predict improvement on a cognitive training task battery, used for patients with schizophrenia, and to determine the proportion of patients whose performance returns to normal following cognitive training

DETAILED DESCRIPTION:
It has been suggested that level of cognitive function is a "rate-limiter" for the efficacy of other psychosocial treatments in schizophrenia. Cognitive remediation, which entails training and practice of successively more difficult cognitive exercises, has shown efficacy in improving cognitive function. However, the rate of improvement has not been uniform among patients receiving this intervention. Given the time- and cost-intensiveness of cognitive remediation, it is important to examine variables that will predict response to this treatment, as well as to examine the clinical significance of any improvement.

The current proposal has two aims: 1) to determine which neuropsychological, demographic, and illness variables predict response to cognitive remediation training; and 2) to determine the proportion of patients whose performance returns to normal following cognitive remediation training. For the first part of the proposed study, 50 outpatients diagnosed with schizophrenia spectrum disorders will be invited to participate in an 8-week trial of cognitive remediation training. Detailed neuropsychological, demographic, symptom and illness course variables will be collected prior to training, at the conclusion of training, and 4 months from study intake. In order to answer the second question, additional data on the computerized task performance for healthy controls will be collected, and compared to patient data, in order to determine what constitutes normal-range performance

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia spectrum disorder
* English speakers
* Clinically stable
* No substance abuse in past 30 days

Exclusion Criteria:

* Traumatic brain injury
* Neurological disease
* Diagnosis of mental retardation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2004-08; Primary Completion 2013-10 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Fiszdon, PhD, Principal Investigator — VA Connecticut Health Care System (West Haven)
Locations (1):
- VA Connecticut Health Care System (West Haven), West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 103 participants were enrolled. Of those, 75 were found eligible, completed baseline assessments and were then randomized to either Arm 1 (n=50) or Arm 2 (n=25). The remaining 28 participants were either discontinued from the study by the PI or chose to withdraw prior to randomization.
Groups:
- Arm 1: cognitive remediation
  cognitive remediation: individual cognitive training
- Arm 2: treatment as usual
Period: Overall Study
Arm/Group | Arm 1 | Arm 2
Started | 50 | 25
Completed | 37 | 18
Not Completed | 13 | 7
Not completed — Withdrawal by Subject | 13 | 7

BASELINE CHARACTERISTICS:
Population: individuals randomized to Arm 1 or Arm 2
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Total
Number analyzed (Participants) | 50 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 25 | 75
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 40 | 16 | 56

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Performance
Description: Change in verbal memory scores from baseline to end of active phase (2 months), measured as trials 1-5 total score on the California Verbal Learning Test -II (range 0-80, higher scores represent better performance).
Time Frame: baseline and 2 months
Population: individuals who were randomized and completed 2 month assessments
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 | Arm 2
Number analyzed (Participants) | 39 | 23
units on a scale | 4.97 (1.38) | -2.30 (1.98)

ADVERSE EVENTS:
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 3/50 | 2/25
Other Adverse Events (participants affected / at risk) | 4/50 | 5/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (N=50) | Arm 2 (N=25)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — participant reported to ER complaining of shortness of breath; determined not to be study related
pulled chest muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — presented to ER with chest pain diagnosed as pulled chest muscle; determined not to be study related
worsening of psychiatric symptoms (Psychiatric disorders) | 1 (1) | 0 (0) — all determined not to be study related
substance abuse (Psychiatric disorders) | 1 (1) | 0 (0) — determined not to be study related
renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — determined not to be study related
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 1 (N=50) | Arm 2 (N=50)
worsening of psychiatric symptoms (Psychiatric disorders) | 2 (2) | 2/25 (2) — determined not to be study related
substance use (Psychiatric disorders) | 0 (0) | 3/25 (3) — determined not to be study related
dizziness (General disorders) | 1 (1) | 0/25 (0) — determined not to be study related
toe pain (Injury, poisoning and procedural complications) | 1 (1) | 0/25 (0) — determined not to be study related

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes